CLINICAL TRIAL: NCT02978274
Title: Natural Killer Cells Reconstitution Kinetics Post T Cells Repleted Haploidentical Transplantation
Brief Title: Natural Killer Cells Reconstitution Kinetics Post Haploidentical Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Professor, Peking University People's Hospital
Other Study IDs: 2016PHB038-01
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Natural Killer Cell Mediated Immunity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PB of patients post transplantation
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- experimental group: MMF withdrawal by engraftment post haplo-SCT
  Interventions: Drug: MMF
- control group: MMF withdrawal by 2 month post haplo-SCT
  Interventions: Drug: MMF

INTERVENTIONS:
Drug: MMF — MMF withdrawal by engraftment post haplo-SCT
  Groups: experimental group
Drug: MMF — MMF withdrawal by 2 month post haplo-SCT
  Groups: control group

SUMMARY:
Patients undergoing haploidentical allo-HSCT will be prospectively enrolled exploring the NK cells phenotype and functional reconstitution.

DETAILED DESCRIPTION:
Patients with hematological malignancies suitable for allo-HSCT but without HLA-identical related or unrelated donors were candidates for the HLA-haploidentical HSCT. Patients undergoing haploidentical allo-HSCT will be prospectively enrolled exploring the NK cells phenotype and functional reconstitution. Peripheral blood will be collected by day15, 30, 60, 90, 180, and 1 year post transplantation.

ELIGIBILITY:
Inclusion Criteria:

* AML or MDS or CML or ALL undergoing haploidentical stem cells transplantation

Exclusion Criteria:

* NR or refractory AML/ALL before transplantation donors from mother or collateral related

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: AML or MDS or CML or ALL undergoing haploidentical stem cells transplantation
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Immune Reconstitution differences between two group | 1 year

SECONDARY OUTCOMES:
Cumulative incidence of Infection differences between two group | 1 year
Cumulative incidence of acute GVHD differences between two group | 100 day
Cumulative incidence of chronic GVHD differences between two group | 1 year
Cumulative incidence of TRM differences between two group | 1 year
Cumulative incidence of relapse differences between two group | 1 year
DFS differences between two group | 1 year
OS differences between two group | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, M.D., PhD, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University Institute of Hematology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao XY, Yu XX, Xu ZL, Cao XH, Huo MR, Zhao XS, Chang YJ, Wang Y, Zhang XH, Xu LP, Liu KY, Huang XJ. Donor and host coexpressing KIR ligands promote NK education after allogeneic hematopoietic stem cell transplantation. Blood Adv. 2019 Dec 23;3(24):4312-4325. doi: 10.1182/bloodadvances.2019000242. PMID 31869417
- [Derived] Kong Y, Wang Y, Zhang YY, Shi MM, Mo XD, Sun YQ, Chang YJ, Xu LP, Zhang XH, Liu KY, Huang XJ. Prophylactic oral NAC reduced poor hematopoietic reconstitution by improving endothelial cells after haploidentical transplantation. Blood Adv. 2019 Apr 23;3(8):1303-1317. doi: 10.1182/bloodadvances.2018029454. PMID 31015207